CLINICAL TRIAL: NCT05366452
Title: Evaluation of the Efficacy of Early Implantation of a Percutaneous Left Ventricular Assist Devices in Acute Coronary Syndrome Complicated by Cardiogenic Shock Compared to Conventional Therapy: a Prospective, Multicenter, Randomized, Controlled and Open-label Clinical Trial
Acronym: ULYSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A02337-32
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPELLA CP GROUP (Experimental): patients will receive IMPELLA CP before PCI on top of conventional therapy based on the same protocol as the control group and emergent culprit PCI
  Interventions: Device: IMPELLA CP
- CONTROL GROUP (Active Comparator): patients will receive IV inotropes associated or not with vasopressors according to the attached protocol and based on the current guidelines (annex 1) (2, 4) in addition to emergent culprit lesion PCI
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Device: IMPELLA CP — Implantation of the IMPELLA CP will be performed using the femoral route in most patients. Echo guided puncture to gain access for IMPELLA CP will be encouraged and a local angiography will be promoted to check the feasibility of device implantation. The implantation will follow gold standard after obtaining an ACT >250 s. As soon as the device is in place it will be started.
  Arms: IMPELLA CP GROUP
Other: Conventional therapy — The patients will receive up to date management according to the consensus of care regarding inotropes and vasopressors in CS (2,4). A dedicated protocol will ensure that management is similar between centers and in both groups. The shock team will be in charge of all therapeutic decisions.
  Arms: CONTROL GROUP

SUMMARY:
The ULYSS study is a randomized, multicenter, interventional and prospective open-label clinical trial. It aims to evaluate the efficacy of the addition of an early IMPELLA CP support on top of optimal medical therapy and culprit lesion PCI compared to optimal medical care and culprit PCI in patients with an ACS complicated by a CS.

A transthoracic echography is required to exclude some non-inclusion criteria as soon as possible and before randomization.

Randomization will be performed after an informed consent is signed by the patient, a family member if he is unable to consent or thanks to the emergent consent procedure if all inclusion criteria are met and there are no non-inclusion criteria. A computer-generated randomization list will be drawn-up using a permuted block design (stratified on center). Each center will have a specific list.

Randomization 1:1 to one of the 2 groups

In all patients, emergent PCI of the culprit lesion will be performed.

* Control group: patients will receive IV inotropes associated or not with vasopressors according to the attached protocol and based on the current guidelines (annex 1) (2, 4) in addition to emergent culprit lesion PCI
* Experimental group: patients will receive IMPELLA CP before PCI on top of conventional therapy based on the same protocol as the control group and emergent culprit PCI

DETAILED DESCRIPTION:
Primary end-point

The primary endpoint (efficacy endpoint) is defined by a composite endpoint assessed at 1 month:

* All cause death;
* Need for ECMO;
* LVAD device implantation;
* Heart transplant

In case of refractory cardiogenic shock (RCS), the use ECMO should be discussed. IMPELLA CP implant is not allowed in the Control group but for venting when required after ECMO implant.

Secondary end-points - Efficacy

At hospital discharge and at one year, the same criteria will be assessed:

* All causes death;
* Need for ECMO;
* Need for LVAD device implantation or for heart transplant

At hospital discharge , at one month and one year, the investigators also want to assess:

* Myocardial infarctions
* Stroke
* Urgent revascularizations (any unplanned revascularization)
* CV deaths
* Procedural success (in-hospital)
* Renal replacement therapies
* Left ventricle ejection fraction at 1 and 12 month follow up
* Quality of life at 1 and 12 months follow up (EQ5D questionnaire).

During hospital stay:

* Durations of catecholamines use
* Length of initial-hospital stay
* Length of stay in intensive care units (ICU + CCU)
* The rate of renal replacement therapies
* Lactates clearance during the first 24 hours
* Area under the curve of CK release during the first 2 days
* Left ventricle ejection fraction at 6 and 12 months follow-up
* Quality of life at one month an one year (EQ5D questionnaire)

Additionally, the investigators will investigated safety and economic criteria of the two strategies.

- Safety

At discharge, at one month and at one year, the investigators will assess:

* The rate of serious adverse events (urgent vascular surgery, transfusion, emboli).
* The rate of BARC bleedings ≥3
* The rate of vascular complications requiring medical or surgical care
* Hemostasis parameters, particularly hemolysis
* Total number of RBC
* Systemic emboli
* Medico-economic the investigators will assess:
* The cost of IMPELLA CP
* The total costs of the intervention
* The EQ5D at baseline and 12 months from PCI (Quality of life through utility health states assessment)
* One year cost-utility analysis: calculated by an incremental cost-utility ratio in terms of costs per additional quality-adjusted life year (QALY).

The rational and methods of the health economic analysis are described in the overall document.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old;
* ACS ≤ 24 hours;
* Cardiogenic shock defined by:
* At least one criteria of low cardiac output defined by
* SBP ≤ 90 mmHg or the need to use inotropes/vasopressors in order to obtain SBP> 90 mmHg
* CI ≤ 2.2L/min/m2
* At least one criteria of left overload defined by
* clinical (killip class ≥ 2),
* biological (NtproBNP > 900pg/ml or BNP > 400pg/ml),
* radiological
* non invasive or invasive hemodynamic evaluation
* At least one criteria of malperfusion defined by
* clinical (marbles, oliguria ≤ 0.5ml/min/kg, cold/clammy skin and extremities,..)
* biological approach (arterial lactate ≥ 2mmol/L, ScVO2 < 60%)
* Stage C or D of the ACC classification of CS
* Revascularization by PCI intended after coronary angiography;
* Lack of significant femoral artery stenosis or other local contra-indication to a 14 Fr sheath;
* Signed informed consent (patient and/or family/relative) or emergency procedure
* Subject affiliated to or beneficiary of a social security system.

Exclusion Criteria:

* Persons referred in articles L.1121-5 to L.1121-8 and L.1122-2 of the Public Health Code:

  * Pregnant, parturient or breastfeeding woman
  * Person deprived of liberty for judicial or administrative decision
  * Adult person under legal protection (any form of public guardianship)
* Onset of shock >24 hours
* CS not related to ACS
* Patient with prolonged cardiac arrest (>5 mins)
* Contra-indications to Impella CP implantations:

  * Isolated right ventricular failure
  * LV thrombus
  * Mechanical aortic valve or heart constrictive device
  * Aortic valve stenosis or calcification (equivalent to an orifice area of 0.6cm2 or less)
  * Moderate to severe aortic insufficiency (echocardiographic assessment graded as ≥ 2)
  * Severe peripheral arterial disease precluding placement of the Impella system
  * Combined cardiorespiratory failure
  * Presence of an Atrial or Ventricular Septal Defect (including post infarctus VSD)
  * Left ventricular rupture Cardiac tamponade
* Mechanical complication of myocardial infarction
* Cerebral deficit with fixed dilated pupils or irreversible neurological pathology
* Anoxic brain injury
* Active bleeding
* Contra-indication to antiplatelet or anticoagulant therapy
* Life expectancy < 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of death from all causes | 1MONTHS
The rate of ECMO placements | 1months
The rate of implementation of the LVAD device | 1 months
The rate of cardiac transplants | 1months

SECONDARY OUTCOMES:
Number of death from all causes | 1 year
The rate of ECMO placements | 1 year
The rate of implementation of the LVAD device | 1 year
The rate of cardiac transplants | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hopitaux De Marseille; LAURENT BONELLO, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, Bouche DU Rhone, France

REFERENCES:
- [Derived] Delmas C, Laine M, Schurtz G, Roubille F, Coste P, Leurent G, Hraiech S, Pankert M, Gonzalo Q, Dabry T, Letocart V, Loubiere S, Resseguier N, Bonello L. Rationale and design of the ULYSS trial: A randomized multicenter evaluation of the efficacy of early Impella CP implantation in acute coronary syndrome complicated by cardiogenic shock. Am Heart J. 2023 Nov;265:203-212. doi: 10.1016/j.ahj.2023.08.066. Epub 2023 Aug 30. PMID 37657594